CLINICAL TRIAL: NCT07317934
Title: A Phase III, Randomized, Open-Label, Active-Controlled Study to Evaluate the Efficacy and Safety of Subretinal Injection of LX102 in Participants With Neovascular Age-Related Macular Degeneration - The STELLAR Trial
Brief Title: Efficacy and Safety of LX102 Gene Therapy in Patients With Neovascular Age-related Macular Degeneration (nAMD) (STELLAR)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innostellar Biotherapeutics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INNOSTELLAR-LX102A03
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Neovascular Age-Related Macular Degeneration (nAMD); Wet AMD
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LX102 (Experimental)
  Interventions: Genetic: LX102
- Aflibercept (Active Comparator)
  Interventions: Biological: Aflibercept

INTERVENTIONS:
Genetic: LX102 — Study eyes will receive a single subretinal injection of LX102.
  Arms: LX102
Biological: Aflibercept — Study eyes will receive 3 monthly loading doses of aflibercetp 2mg IVT and aflibercept 2mg IVT every 8 weeks.
  Arms: Aflibercept

SUMMARY:
This is a Phase III, randomized, open-label, active-controlled study to evaluate the efficacy and safety of subretinal injection of LX102 in participants with neovascular age-related macular degeneration. The study will evaluate a single subretinal injection of LX102 compared to an active comparator. The primary endpoint of this study is the mean change from D0 in BCVA based on an average at weeks 40 and 48.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written, signed informed consent for this study;
2. Age ≥50 and ≤80 years old;
3. active CNV secondary to nAMD in the study eye confirmed by FFA or OCT;
4. The BCVA between 24 and 78 letters (inclusive) in the study eye at Screening;
5. Demonstrated clinical response to aflibercept treatments in the study eye confirmed by the Reading Center;
6. No anti-VEGF therapy in study eye within 28 days before screening;
7. Must be pseudophakic in the study eye (at least 4 weeks after cataract surgery).

Exclusion Criteria:

1. Any condition in the investigator's opinion that could limit VA improvement in the study eye.
2. CNV or macular edema in the study eye secondary to any causes other than AMD
3. Subfoveal fibrosis or atrophy in the study eye, as determined by CRC;
4. History of retinal detachment in the study eye at any time;
5. History of idiopathic or autoimmune uveitis in either eye;
6. Advanced glaucoma in the study eye;
7. History of vitrectomy surgery in the study eye;
8. History of intraocular surgery within 1 month before screening in the study eye;
9. History of ocular or systemic gene therapy;
10. Recent myocardial infarction, cerebrovascular accident, or transient ischemic attack within the past 6 months.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2032-06-04 (Estimated)

PRIMARY OUTCOMES:
Mean change from D0 in BCVA based on an average at weeks 40 and 48. | Weeks 40 and 48
  Mean change from D0 in BCVA as measured by the early treatment diabetic retinopathy study (ETDRS) visual acuity chart based on an average at weeks 40 and 48.

SECONDARY OUTCOMES:
Proportion of participants with improved BCVA | Week 48
  Proportion of participants with improved BCVA at week 48
Proportion of participants with worsened BCVA | Week 48
  Proportion of participants with worsened BCVA at week 48
Mean change from D0 in CST based on an average at weeks 40 and 48 | Weeks 40 and 48
  Mean change from D0 in central subfield thickness (CST) based on an average at weeks 40 and 48
Proportion of participants without SRF/IRF on OCT at week 48 | Week 48
  Proportion of participants without SRF/IRF on OCT at week 48
Proportion of participants who were supplemental anti-VEGF injection-free | Through 48 weeks
  Proportion of participants with no supplemental anti-VEGF injection through 48 weeks
Proportion of participants who received 1 or 2 aflibercept injections | Through 48 weeks
  Proportion of participants received ≤2 supplemental anti-VEGF injections through 48 weeks
Supplemental anti-VEGF injection annualized rate after LX102 administration through Week 48 | Through 48 weeks
  Mean annualized number of anti-VEGF injections after LX102 administration through 48 weeks.
Incidence of ocular and nonocular AEs and SAEs | 48 weeks
  Incidence of Adverse events (AE) and Serious adverse events (SAE) over 48 weeks
Immunogenicity characteristics of LX102 | 48 weeks
  Immunogenicity measurements (LX102 randomized participants) ; measure description: Immunogenicity measurements (vector shedding, serum antibodies to AAV2 and serum antibodies to LX102 TP)

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Joint Shantou International Eye Center, Shantou University and the Chinese University of Hong Kong, Shantou, Guangdong
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Zhongshan, Guangdong
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Central Theater Command General Hospital of PLA, Wuhan, Hubei
  - The Second Xiangya Hospital, Central South University, Changsha, Hunan
  - Aier Eye Hospital Group Co., LTD. Changsha Aier Eye Hospital, Changsha, Hunan
  - The Affiliated Eye Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Xuzhou First People's Hospital, Xuzhou, Jiangsu
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Eye Hospital, Jinan, Shandong
  - Qingdao Eye Hospital Affiliated to Shandong First Medical University, Qingdao, Shandong
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Xinhua Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Eye Hospital, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Xi 'an People's Hospital (Xi 'an No.4 Hospital), Xi’an, Shanxi
  - The First Affiliated Hospital of Air Force Medical University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Eye Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The Eye Hospital of Wenzhou Medical University, Wenzhou, Zhejiang